CLINICAL TRIAL: NCT06972563
Title: The Effect of Psychoeducation Based on Acceptance and Commitment Therapy Applied to Patients Diagnosed With Generalized Anxiety Disorder on Cognitive Avoidance Levels and Coping Attitudes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arzu Çalışkan (Other)
Responsible Party: Sponsor-Investigator, Arzu Çalışkan, Nurse, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Gaziantep Üniversitesi
Record Dates: First submitted 2024-09-25; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Acceptance and Commitment Therapy; Cognitive Avoidance; Coping Attitudes
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Psychoeducation Based on Acceptance and Commitment Therapy Applied to Patients Diagnosed with Generalized Anxiety Disorder
  Interventions: Other: Psychoeducation Based on Acceptance and Commitment Therapy Applied to Patients Diagnosed with Generalized Anxiety Disorder
- Control (Other): The initiative was not implemented.
  Interventions: Other: The initiative was not implemented.

INTERVENTIONS:
Other: Psychoeducation Based on Acceptance and Commitment Therapy Applied to Patients Diagnosed with Generalized Anxiety Disorder — Psychoeducation Based on Acceptance and Commitment Therapy Applied to Patients Diagnosed with Generalized Anxiety Disorder
  Arms: Experiment
Other: The initiative was not implemented. — The initiative was not implemented.
  Arms: Control

SUMMARY:
This study will be conducted to determine the effects of acceptance and commitment therapy-based psychoeducation on cognitive avoidance levels and coping attitudes in patients diagnosed with generalized anxiety disorder.

H0: Acceptance and commitment therapy-based psychoeducation has no effect on the cognitive avoidance levels and coping attitudes of patients diagnosed with generalized anxiety disorder.

H1: Acceptance and commitment therapy-based psychoeducation reduces the cognitive avoidance levels of patients diagnosed with generalized anxiety disorder.

H2: Acceptance and commitment therapy-based psychoeducation affects the coping attitudes of patients diagnosed with generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with generalized anxiety disorder according to DSM-5 diagnostic criteria and receiving outpatient treatment
* Being literate
* Having no problems understanding or speaking Turkish
* Being in the 18-65 age group
* Having not received such training in the last 6 months

Exclusion Criteria:

* Those diagnosed with another comorbid mental illness Patients with a mental condition that makes cooperation impossible, such as intellectual disability or memory impairment
* The illiterate
* Patients who do not consent to be interviewed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Measuring the effect of cognitive avoidance levels of patients diagnosed with generalized anxiety disorder | 1 month
  Patients answered cognitive avoidance scale. Cognitive Avoidance Scale (Cope) measures cognitive avoidance strategies. COA is a self-assessment type scale. The five (1-5) point Likert-type scale (1-strongly disagree, 5-strongly agree) measures 25 items of COA. The score that can be obtained from the scale is between 12 and 125. In order to calculate the total score, it is necessary to sum the answers given to all items. A high score indicates that a cognitive avoidance strategy is used in the face of problems.

SECONDARY OUTCOMES:
coping attitudes of patients diagnosed with generalized anxiety disorder | 1 month
  The scale is a 4-point Likert-type scale. When scoring the items, 1 point is given for "I Never Do This", 2 points for "I Rarely Do This", 3 points for "I Do This" and 4 points for "I Often Do This". There are no negative items in the scale. The highest score that can be obtained from the scale is 160, the lowest score is 40. A high score obtained from the scale means a high level of coping attitude, and a low score means a low level of coping attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Eğitim ve Araştırma Hastanesi, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No detailed permission was obtained from the owners of the collected data.